CLINICAL TRIAL: NCT01099774
Title: Safety and Efficacy of Different Formulations of Bimatoprost Ophthalmic Solution in Patients With Glaucoma or Ocular Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 192024-048
Record Dates: First submitted 2010-04-06; First posted 2010-04-08 (Estimated); Results first posted 2012-04-27 (Estimated); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Glaucoma; Ocular Hypertension
MeSH Terms: conditions — Glaucoma; Ocular Hypertension | interventions — Bimatoprost; Ophthalmic Solutions

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bimatoprost 0.03% Formulation B Ophthalmic Solution (Experimental): Bimatoprost 0.03% Formulation B Ophthalmic Solution
  Interventions: Drug: Bimatoprost 0.03% Formulation B Ophthalmic Solution
- Bimatoprost 0.03% Ophthalmic Solution (Active Comparator): Bimatoprost 0.03% Ophthalmic Solution
  Interventions: Drug: Bimatoprost 0.03% Ophthalmic Solution

INTERVENTIONS:
Drug: Bimatoprost 0.03% Formulation B Ophthalmic Solution — One drop administered in each eye, every evening, for 12 weeks
  Arms: Bimatoprost 0.03% Formulation B Ophthalmic Solution
Drug: Bimatoprost 0.03% Ophthalmic Solution — One drop administered in each eye, every evening, for 12 weeks
  Other Names: LUMIGAN®
  Arms: Bimatoprost 0.03% Ophthalmic Solution

SUMMARY:
This study will evaluate the safety and efficacy of bimatoprost 0.03% formulation B ophthalmic solution with LUMIGAN® (bimatoprost ophthalmic solution 0.03%) once daily for 12 weeks in patients with glaucoma or ocular hypertension

ELIGIBILITY:
Inclusion Criteria:

* Patient has ocular hypertension or glaucoma in both eyes
* Requires IOP-lowering therapy in each eye

Exclusion Criteria:

* Active or recurrent eye disease that would interfere with interpretation of study data in either eye
* History of any eye surgery or laser in either eye within 6 months
* Required chronic use of other eye medications during the study
* Anticipated wearing of contact lenses during the study.
* Intermittent use of oral, intramuscular, or intravenous corticosteroids within 21 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 597 (Actual)
Dates: Start 2010-05-01 (Actual); Primary Completion 2011-04-29 (Actual); Study Completion 2011-04-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (1):
- Newport Beach, California, United States

REFERENCES:
- [Background] Day DG, Walters TR, Schwartz GF, Mundorf TK, Liu C, Schiffman RM, Bejanian M. Bimatoprost 0.03% preservative-free ophthalmic solution versus bimatoprost 0.03% ophthalmic solution (Lumigan) for glaucoma or ocular hypertension: a 12-week, randomised, double-masked trial. Br J Ophthalmol. 2013 Aug;97(8):989-93. doi: 10.1136/bjophthalmol-2012-303040. Epub 2013 Jun 6. PMID 23743437

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Bimatoprost 0.03% Formulation B Ophthalmic Solution | Bimatoprost 0.03% Ophthalmic Solution
Started | 302 | 295
Completed | 296 | 289
Not Completed | 6 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bimatoprost 0.03% Formulation B Ophthalmic Solution | Bimatoprost 0.03% Ophthalmic Solution | Total
Number analyzed (Participants) | 302 | 295 | 597
Age, Customized [Number; unit: Participants]
  <45 years | 8 | 11 | 19
  Between 45 and 65 years | 159 | 134 | 293
  >65 years | 135 | 150 | 285
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 170 | 181 | 351
  Male | 132 | 114 | 246

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Worse Eye Intraocular Pressure (IOP) at Week 12
Description: Change from baseline in worse eye IOP at Week 12 . IOP is a measurement of fluid pressure inside the eye. IOP measurements in the worse eye were evaluated at hours 0, 2, and 8. A negative number change from baseline indicated a reduction in IOP, and a positive number change from baseline indicated an increase in IOP.
Time Frame: Baseline, Week 12
Population: Per Protocol Population: All randomized patients who did not have a protocol violation that significantly affected the conduct or the results of the trial.
Measure: Mean (Standard Deviation); unit: Millimeters of Mercury (mmHg)
Arm/Group | Bimatoprost 0.03% Formulation B Ophthalmic Solution | Bimatoprost 0.03% Ophthalmic Solution
Number analyzed (Participants) | 295 | 291
Millimeters of Mercury (mmHg)
  Baseline Hour 0 | 24.90 (2.364) | 24.86 (2.161)
  Baseline Hour 2 | 23.79 (2.992) | 23.78 (2.753)
  Baseline Hour 8 | 22.81 (3.168) | 22.80 (3.301)
  Change from Baseline Hour 0 at Week 12 | -7.49 (2.900) | -7.77 (3.029)
  Change from Baseline Hour 2 at Week 12 | -7.06 (3.333) | -7.11 (3.192)
  Change from Baseline Hour 8 at Week 12 | -5.93 (3.432) | -6.06 (3.602)

2. Primary Outcome: Average Eye IOP at Week 12
Description: Average Eye IOP at Week 12 . IOP is a measurement of fluid pressure inside the eye. IOP measurements were evaluated at hours 0, 2, and 8 in both eyes and the average IOP of both eyes at each time point were reported. Baseline data are included for reference only.
Time Frame: Baseline, Week 12
Population: Intent to Treat Population: all randomized patients.
Measure: Mean (Standard Deviation); unit: Millimeters of Mercury (mmHg)
Arm/Group | Bimatoprost 0.03% Formulation B Ophthalmic Solution | Bimatoprost 0.03% Ophthalmic Solution
Number analyzed (Participants) | 302 | 295
Millimeters of Mercury (mmHg)
  Baseline Hour 0 | 24.53 (2.196) | 24.46 (2.019)
  Baseline Hour 2 | 23.30 (2.848) | 23.26 (2.613)
  Baseline Hour 8 | 22.31 (2.974) | 22.29 (3.110)
  Week 12 Hour 0 | 17.25 (2.804) | 16.96 (2.886)
  Week 12 Hour 2 | 16.51 (2.900) | 16.55 (2.863)
  Week 12 Hour 8 | 16.64 (2.820) | 16.59 (2.735)

3. Primary Outcome: Average Eye IOP at Week 6
Description: Average Eye IOP at Week 6 . IOP is a measurement of fluid pressure inside the eye. IOP measurements were evaluated at hours 0, 2, and 8 in both eyes and the average IOP of both eyes at each time point were reported.
Time Frame: Week 6
Population: Intent to Treat Population: all randomized patients.
Measure: Mean (Standard Deviation); unit: Millimeters of Mercury (mmHg)
Arm/Group | Bimatoprost 0.03% Formulation B Ophthalmic Solution | Bimatoprost 0.03% Ophthalmic Solution
Number analyzed (Participants) | 302 | 295
Millimeters of Mercury (mmHg)
  Week 6 Hour 0 | 17.16 (2.967) | 17.08 (2.957)
  Week 6 Hour 2 | 16.52 (2.855) | 16.45 (2.766)
  Week 6 Hour 8 | 16.56 (2.838) | 16.32 (2.702)

4. Primary Outcome: Average Eye IOP at Week 2
Description: Average Eye IOP at Week 2 . IOP is a measurement of fluid pressure inside the eye. IOP measurements were evaluated at hours 0, 2, and 8 in both eyes and the average IOP of both eyes at each time point were reported.
Time Frame: Week 2
Population: Intent to Treat Population: all randomized patients.
Measure: Mean (Standard Deviation); unit: Millimeters of Mercury (mmHg)
Arm/Group | Bimatoprost 0.03% Formulation B Ophthalmic Solution | Bimatoprost 0.03% Ophthalmic Solution
Number analyzed (Participants) | 302 | 295
Millimeters of Mercury (mmHg)
  Week 2 Hour 0 | 17.40 (2.732) | 17.14 (2.677)
  Week 2 Hour 2 | 16.68 (2.759) | 16.43 (2.581)
  Week 2 Hour 8 | 16.61 (2.766) | 16.39 (2.795)

ADVERSE EVENTS:
Arm/Group | Bimatoprost 0.03% Formulation B Ophthalmic Solution | Bimatoprost 0.03% Ophthalmic Solution
Serious Adverse Events (participants affected / at risk) | 2/301 | 5/295
Other Adverse Events (participants affected / at risk) | 72/301 | 77/295
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bimatoprost 0.03% Formulation B Ophthalmic Solution (N=301) | Bimatoprost 0.03% Ophthalmic Solution (N=295)
Ovarian Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Spinal Compression Fracture (Injury, poisoning and procedural complications) | 1 | 0
Atrial Fibrillation (Cardiac disorders) | 0 | 1
Convulsion (Nervous system disorders) | 0 | 1
Death (General disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
Transitional Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bimatoprost 0.03% Formulation B Ophthalmic Solution (N=301) | Bimatoprost 0.03% Ophthalmic Solution (N=295)
Conjunctival Hyperaemia (Eye disorders) | 72 | 77

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo